CLINICAL TRIAL: NCT03414619
Title: The Role of Cognitive Control in the Transdiagnostic Conceptualization of "Intrusive Thoughts"
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Health Resources in Action, Inc. (Other)
Responsible Party: Principal Investigator, Ryan Jane Jacoby, Ryan Jane Jacoby, Ph.D., Clinical Psychologist, OCD and Related Disorders Program, Massachusetts General Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017P002114
Record Dates: First submitted 2018-01-23; First posted 2018-01-30 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Major Depressive Disorder
Keywords: OCD; GAD; MDD; Rumination; Obsession; Worry
MeSH Terms: conditions — Obsessive-Compulsive Disorder; Generalized Anxiety Disorder; Depressive Disorder, Major; Rumination Syndrome; Obsessive Behavior

STUDY DESIGN:
Intervention Model Description: The current study has two diagnostic arms (the Intrusive Thoughts group and the Non-Psychiatric Control group) all receiving a single interventional protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intrusive Thoughts Group (Experimental): Clinically significant intrusive thought in the domain of obsessions, worries, or depressive ruminations with a score above the clinical mean (≥ 37) on the trait repetitive negative thinking measure (Perseverative Thinking Questionnaire, PTQ). These participants will receive the Cognitive Control Tasks and Script Driven Imagery Intervention.
  Interventions: Behavioral: Cognitive Control Tasks and Script Driven Imagery
- Non-psychiatric Control Group (Experimental): A score 1 SD below the community mean (≤ 15) on the trait repetitive negative thinking measure (Perseverative Thinking Questionnaire, PTQ). These participants will also receive the Cognitive Control Tasks and Script Driven Imagery Intervention.
  Interventions: Behavioral: Cognitive Control Tasks and Script Driven Imagery

INTERVENTIONS:
Behavioral: Cognitive Control Tasks and Script Driven Imagery — All participants will receive a structured diagnostic assessment and complete self-report questionnaires about cognitive factors and anxiety/mood symptoms. They then will complete a battery of neuropsychological executive functioning tasks on the computer, each of which measures a different facet of cognitive control (i.e., response inhibition, cognitive flexibility, and attentional control). Finally, they will be guided through a standardized script-driven imagery paradigm that involves generating and listening to an individualized imaginal script associated with a moderately distressing intrusive thought. Self-report and psychophysiological data will be collected during this exercise.

SUMMARY:
The investigators are examining whether difficulties with cognitive control (i.e., the ability to stop one's thought process and shift attention) is a common problem across three types of repetitive, negative thinking: obsessions (as seen in obsessive compulsive disorder, OCD), worries (as seen in generalized anxiety disorder, GAD), and ruminations (as seen in major depressive disorder, MDD).

DETAILED DESCRIPTION:
The primary aims of this study are to utilize self-report and behavioral measures to examine whether cognitive control is a common factor across three types of repetitive negative thinking (RNT): obsessions in OCD, worries in GAD, and ruminations in MDD. Specifically, the investigators aim to test whether individuals with obsessions, worries, and depressive ruminations demonstrate impaired cognitive control on executive functioning neuropsychological tasks (i.e., response inhibition, set shifting, attentional disengagement) relative to individuals without any psychiatric diagnoses. Additionally, the investigators will examine whether these deficits are associated with self-report measures of RNT as well as in vivo responding during a laboratory paradigm designed to induce intrusive thinking. Findings could inform psychological treatment of these problematic intrusions using novel transdiagnostic approaches.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age 18+)
2. Intrusive thoughts group: Clinically significant intrusive thought in the domain of obsessions, worries, or depressive ruminations with a score above the clinical mean (≥ 37) on the trait repetitive negative thinking measure (Perseverative Thinking Questionnaire, PTQ)
3. Non-psychiatric control (NPC) group: A score 1 SD below the community mean (≤ 15) on the trait repetitive negative thinking measure (PTQ)
4. Sufficient fluency of English to understand study procedures and questionnaires
5. Ability to provide informed consent.
6. Comfortable and capable of using a computer and completing reaction-time tasks.

Exclusion Criteria:

1. Acute psychosis, mania, or suicidality
2. Diagnosis of post-traumatic stress disorder (PTSD; in order to preserve diagnostic clarity of the domains of intrusive thoughts under investigation)
3. Serious neurological disorder or impairment (e.g., brain damage, blindness), attention deficit hyperactivity disorder (ADHD), intellectual disability, or autism.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2018-05-18 (Actual); Primary Completion 2020-03-06 (Actual); Study Completion 2020-03-06 (Actual)

PRIMARY OUTCOMES:
Commission Errors on the Go/No Go Task | Day 1
  In the Go/No Go Task participants press a button immediately upon detecting a target stimulus (e.g., a square), but are told to refrain from responding to a "no go" stimulus (e.g., a cross of similar size). The main outcome is commission errors (i.e., responding to a "no go" stimulus).
Response time on the Stroop Color Word Test | Day 1
  In the Stroop Color Word Test participants are asked to name the color of the ink in which words are printed, rather than reading the words.
Perseverative Errors on the Wisconsin Card Sort Test | Day 1
  In the Wisconsin Card Sort Test participants are asked to match a stack of response cards to four stimulus cards without knowing the matching rule. They receive feedback for each trial about whether their matching was correct or not. After ten consecutive correct trials, the matching criterion changes without notice requiring the use of flexible goal-driven strategies.
Gaze latency on the Attentional Engagement-Disengagement Task | Day 1
  In the Attentional Engagement-Disengagement Task two emotional facial stimuli are presented on the computer screen (i.e., happy, disgusted, fearful, and sad faces paired with neutral faces) and eye tracking (when participants shift from the emotional to neutral face and vice versa) is measured.

SECONDARY OUTCOMES:
Perseverative Thinking Questionnaire (PTQ) | Day 1
  The Perseverative Thinking Questionnaire is a 15-item measure of repetitive, negative thinking considered independent of disorder-specific content (e.g., "The same thoughts keep going through my mind again and again").
State measure of intrusive thinking | Day 1
  Participants will be asked questions on a visual analog scale from 0 "not at all" to 100 "extremely" regarding state experiences of intrusive thoughts.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Jacoby, Ph.D., Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Daniel KE, Wilhelm S, Jacoby RJ. Predictors of polyregulation and its effectiveness following exposure to One's most personally distressing intrusive thought. J Behav Ther Exp Psychiatry. 2025 Mar;86:102001. doi: 10.1016/j.jbtep.2024.102001. Epub 2024 Dec 1. PMID 39626971